CLINICAL TRIAL: NCT02653651
Title: A Comparison Between the Effects of Perioperative Intravenous Lidocaine and Ketamine on Acute and Chronic Pain After Open Nephrectomy: A Prospective, Double-blind, Randomized, Placebo Controlled Study
Brief Title: Effects of Perioperative Intravenous Lidocaine and Ketamine on Acute and Chronic Pain After Open Nephrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ali JENDOUBI, MD, Assistant Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UTuniselmanar
Record Dates: First submitted 2016-01-01; First posted 2016-01-12 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Postoperative Pain
Keywords: Ketamine; Lidocaine; Nephrectomy; Chronic pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Ketamine; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketamine (Active Comparator): Ketamine infused at 0.1 mg/kg/hour
  Interventions: Drug: Ketamine
- Lidocaine (Experimental): Lidocaine infused at 1 mg/kg/hour
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): An equal volume of saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine infused at 0.1 mg/kg/hour
  Arms: Ketamine
Drug: Lidocaine — Lidocaine infused at 1 mg/kg/hour
  Arms: Lidocaine
Drug: Placebo — An equal volume of saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Open nephrectomy is one of the most common surgical procedures in urologic practice. Pain after surgery remains a significant clinical problem as it impairs recovery adversely and may lead to the transition to chronic pain. The open approach represents a major physical trauma including postoperative pain and discomfort in the convalescence period. Adequate control of postoperative pain facilitates earlier mobilization and rehabilitation. Patient-controlled analgesia (PCA) is effective to treat pain at rest, but seems to be inadequate for dynamic analgesia and may also elicit side effects that may delay hospital discharge. Preventing early and late postsurgical pain is an important challenge for anesthesiologists and surgeons.

Ketamine (N-Methyl-D-Aspartate receptor antagonist) and lidocaine (sodium channel blocker) are popular analgesic adjuvants for improving perioperative pain management. The investigators designed this double-blind, placebo controlled study to test and compare the preventive effects of perioperative intravenous ketamine and lidocaine on early and chronic pain after elective open nephrectomy.

The investigators propose a double-blind placebo-controlled study of patients undergoing elective open nephrectomy. All patients will receive normal "patient-controlled analgesia morphine" in addition to study drugs or placebo. Research will be conducted at Charles Nicolle teaching hospital.

DETAILED DESCRIPTION:
Participants will be randomized into one of three study groups: Group L: intravenous lidocaine: bolus of 1.5 mg/kg at induction of anesthesia followed by infusion of 1 mg/kg/h intraoperatively and for 24 h postoperatively. Group K: Ketamine: bolus of 0.15 mg/kg followed by infusion of 0.1 mg/kg/h intraoperatively and for 24 h postoperatively. Control Group C: an equal volume of saline. The anesthetic technique will be standardized, and the postoperative assessments included pain scores, opioid consumption, recovery of bowel function and 6-minute walk distance (6-MWD) on the fourth postoperative morning. At 3 months, patients will be questioned for chronic postoperative pain using the Neuropathic Pain 4 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>/=18)
2. male or female
3. Undergoing elective open nephrectomy
4. General anesthesia
5. Subject is American Society of Anesthesiologists (ASA) physical status 1 or 2.

Exclusion Criteria:

1. Pregnancy and breastfeeding
2. Cognitively impaired (by history)
3. Subject with a history of psychosis
4. Subject known to have significant hepatic disease
5. History of previous cardiac arrhythmia
6. Subject for whom opioids or ketamine are contraindicated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | 24 hours
  the total amount of morphine consumed during follow up period

SECONDARY OUTCOMES:
Postoperative nausea and vomiting using a Verbal Rating Scale | 48 hours
  Investigators will ask patients to grade the severity of their nausea and vomiting episodes using a verbal rating scale
Functional recovery assessed by 6 minute walk test (6MWT) | the fourth postoperative morning
chronic postoperative pain assessed by the Neuropathic Pain 4 questionnaire. (NP4) | At 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali JENDOUBI, Principal Investigator — University Tunis El Manar
Locations (1):
- Ali JENDOUBI, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No